CLINICAL TRIAL: NCT05308368
Title: Analysis and Suppression of Tremor During Grasp Using Ultrasound Imaging and Electrical Stimulation
Acronym: Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Nitin Sharma, Associate Professor, North Carolina State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19247; 5R21EB032059 (NIH)
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor | interventions — Ultrasonography; Electromyography

STUDY DESIGN:
Intervention Model Description: The central objective of this study is to collect experimental data to develop tremor models and suppression methods and validate these methods on participants with tremor.
  This study is performed with two sets of subjects: people with Parkinson's Disease and Essential Tremor and people without any neurological disorders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tremor Group (Experimental): Individuals with either parkinson's disease or essential tremor will be recruited in this group
  Interventions: Device: Ultrasound Imaging; Device: Electromyography; Device: Inertial Measurement Units (IMU); Device: Functional Electrical Stimulation (FES)
- Able Body Group (Experimental): Individuals with no disorders will be recruited in this group
  Interventions: Device: Ultrasound Imaging; Device: Electromyography; Device: Inertial Measurement Units (IMU); Device: Functional Electrical Stimulation (FES)

INTERVENTIONS:
Device: Ultrasound Imaging — We will collect ultrasound images during the grasping motion for both groups
Device: Electromyography — We will collect electromyography (EMG) signals of both the flexor and extensor muscles of the wrist during the grasping motion for both groups
Device: Inertial Measurement Units (IMU) — We will use data from the ultrasound images and EMG to develop a tremor model. The model will be validated in comparison to joint angle measurements from an Inertial Measurement Unit (IMU) collected during the grasping motion
Device: Functional Electrical Stimulation (FES) — We will use the develop closed-loop control methods for tremor suppression using information from the ultrasound-image based tremor models. FES will be used to provide stimulation that will help with tremor suppression

SUMMARY:
Individuals experiencing tremors face difficulty performing activities of daily living caused by involuntary oscillation of the muscles in the hands and arms. Current solutions to help suppress tremors include medication, surgery, assistive devices and lifestyle change. However, each of these has a drawback of its own including cost and unwanted side effects. Aside from the solutions listed, it has been shown that functional electrical stimulation (FES) is a possible solution to help suppress tremor. Additionally, FES can be combined with different technologies including accelerometers, gyroscopes and motion capture to develop a closed loop system for tremor suppression. However, this has drawbacks including signal interference and the need for multiple sensor to fully classify the tremor. Ultrasound imaging solves some of these issues because it can provide a direct visualization of hand muscles that contribute to tremor. This study will focus on detecting characterizing and differentiating tremors from voluntary hand motion using ultrasound imaging. The results obtained from this study will help design FES-based tremor-suppression techniques in the future. This study will target both subjects with different tremor disorders and able bodied subjects.

ELIGIBILITY:
Inclusion Criteria (Tremor Group):

1. At least 40 years of age, and no more than 90 years of age.
2. Meet UK Parkinson's disease brain bank diagnostic criteria
3. Have clinical evidence of rest tremor of one or both upper extremities defined as involuntary, rhythmic oscillations about any joint within the upper extremities
4. Tremor amplitude must be at minimum 1 cm as determined by expert opinion by a movement disorders specialist.
5. Due to the nature of measurements occurring during a grasp maneuver, the tremor must be deemed to become re-emergent with a fixed posture. This shall be defined by development of postural tremor that does not begin immediately upon grasping the vertical object, but instead with a delay in development of oscillatory movement of at least half a second as timed by a stopwatch, and that may grow in amplitude over seconds to maximum amplitude without changing the force of the grasp at first. Note that within-individual intermittency and variability of tremor can be influenced by anxiety, stress, cold temperature, and fatigue. In an effort to reduce this variability, we will have subjects perform tasks in a comfortable area, providing up to 20 minutes to allow them to relax in a temperature-neutral location, and reduce anxiety

Exclusion Criteria (Tremor Group):

1. Muscle weakness as determined by Medical Research Council grade less than 5/5 on direct testing in the upper limb afflicted with rest tremor
2. Infection at the upper limb at time of assessment
3. Pre-existing, concomitant neuromuscular or cerebellar disorders
4. Use of medications that can alter the function of the neuromuscular junction.
5. Those with concomitant essential tremor as determined by history or confirmed by movement disorders specialist prior to assessments.

Inclusion Criteria (Able Body):

Subjects will fall under the able body category if they exhibit no movement disorders and can perform grasping motion with no inhibition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Engineering Building III, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of this research group. However, selected data may be published in academic journals, conference papers, or other publications. This data will be de-identified, and will not include the full set of data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2021-recruitment of 1 participant 2022- recruitment of 8 participants 2023- recruitment of 3 participants
Period: Overall Study
Arm/Group | Tremor Group
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study's objective was to quantify the suppression effects of afferent peripheral nerve stimulation and measure tremor frequency through new sensing approaches in people with Essential Tremor or Parkinson's disease. Another objective was to model tremor dynamics through data-driven approaches. Since the able-bodied group does not exhibit tremor, they were not recruited for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tremor Group | Able Body Group | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 8 |  | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 8 |  | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 12 |  | 12
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 1 |  | 1
  Black or African American | 0 |  | 0
  White | 11 |  | 11
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Tremor Model Accuracy
Description: The investigators will use ultrasound features collected on participants to develop novel models for tremor that can accurately predict the joint position. The joint position measured by the IMU will used as a benchmark and the root mean squared error (RMSE [Deg.]) between the model's predicted joint angle and the true angle will be used as a metric. A higher RMSE (in the scale of 0-100%) implies lower model accuracy.
Time Frame: Through Completion of Study, an average of 3 years
Population: Only participants who completed assessment are included.
Measure: Mean (Standard Deviation); unit: Normalized RMSE (%)
Arm/Group | Tremor Group
Number analyzed (Participants) | 6
Normalized RMSE (%)
  Tremor Model Prediction Accuracy without stimulation | 24 (4.49)
  Tremor Model Prediction Accuracy with stimulation | 21 (2.66)

2. Primary Outcome: Ultrasound Imaging Based Frequency Detection
Description: The investigators will benchmark the performance of the ultrasound features (fascicle length [mm], muscle thickness [mm]) in detecting the actual tremor frequency (Hz) measured by an inertial measurement unit (IMU) sensor and electromyography (EMG). Here error between the tremor frequency measured with IMU and the ultrasound feature-derived tremor frequency is reported. A lower mean error (0-100%) implies higher concurrence with the IMU-derived or EMG-derived tremor frequency.
Time Frame: Through Completion of Study, an average of 3 years
Population: Only participants who completed assessment are included in the analysis
Measure: Mean (Standard Deviation); unit: Error percentage (%)
Arm/Group | Tremor Group
Number analyzed (Participants) | 6
Error percentage (%)
  Frequency Comparison with IMU | 8.9 (0.57)
  Frequency Comparison with EMG | 6.4 (0.39)

3. Primary Outcome: Tremor Suppression (Percentage)
Description: The investigators will use the developed tremor models to develop closed loop control methods using FES which enable tremor suppression. The goal of the controller will be to maintain a desired wrist angle position while performing a grasping motion. A tremor suppression ratio metric, formulated as 1-(W_t/W_b), where W_t is the angular velocity of the wrist around the vertical during periods in which stimulation was turned on and W_b is the angular velocity during baseline periods without any stimulation, is used as an evaluation metric. A higher tremor suppression ratio (0-100%) means higher effectiveness in suppressing the tremor.
Time Frame: Through Completion of Study, an average of 3 years
Population: Only participants who completed these experiments are included in the analysis
Measure: Mean (Standard Deviation); unit: Percentage Suppression
Arm/Group | Tremor Group
Number analyzed (Participants) | 8
Percentage Suppression | 62.4 (18.93)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Tremor Group
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT05308368/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05308368/SAP_001.pdf